CLINICAL TRIAL: NCT06612827
Title: Development of Tumor Organoids From Undifferentiated Primary Carcinomas to Guide Therapeutic Decisions
Acronym: OCAPI
Status: Recruiting | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A01326-41
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Undifferentiated Carcinoma
Keywords: tumoroid; organoid
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood and tumor collection: Blood and tumor collection before treatment initiation
  Interventions: Other: organoid etablishment

INTERVENTIONS:
Other: organoid etablishment — Prior to initiation of 1st-line therapy:
  * Collection of an additional study-specific tumor sample for tumoroid analysis (1 fresh tumor sample)
  * A blood test blood a for tumoroid realization and :
  * Analysis of ex vivo tumoroid response to treatment and correlation with patient response in vivo
  * Analysis of correlation between in vivo and ex vivo tumor characteristics
  * Analysis of first- and second-line survival rates and overall survival

SUMMARY:
The study is based on the constitution of a collection of tumor and blood samples for the development of tumoroid for functional tests to predict clinical response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with undifferentiated primary carcinoma (UPC) with histological and immunohistochemical evidence, validated in a local and/or national UPC multidisciplinary consultation
* Patient with indication for systemic 1st-line treatment at the time of inclusion. Treatment may already have begun at the time of inclusion, but within the limit of 2 treatment cycles administered.
* Patient with life expectancy greater than 3 months
* Patient of legal age
* Patient affiliated to a social security scheme
* Signature of informed consent prior to any specific study procedure

Exclusion Criteria:

* Persons deprived of their liberty or under guardianship (including curatorship)
* Pregnant or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with undifferentiated primary carcinoma (UPC) with indication for 1st-line treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2032-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of establishment of exploitable tumor organoids | through study completion, an average of 3 years
  Rate of establishment usable tumor organoids for predictive tests of response to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided